CLINICAL TRIAL: NCT01945892
Title: Ozurdex as an Treatment Option for Macula Edema Due to Irvine Gass Syndrome
Brief Title: Dexamethasone-Implant for the Treatment of Macula Edema Due to Irvine Gass Syndrome
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Wolfgang Mayer, Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: MAF/ISS/OPH/RET/011
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Macular Edema; Visual Acuity
Keywords: macular edema, irvine gass syndrome, ozurdex
MeSH Terms: conditions — Macular Edema | interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Irvine Gass Syndrome: Patients older than 18 years who develop macula edema secondary to cataract surgery.
  Group may receive intravitreal Ozurdex medication in case of persistent macular edema.
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — - Consent agreement - Patients should be informed that it is possible to get an active medication (Ozurdex implant) as an "on label" indication from the health insurance company if the diagnosis is accepted as an intraocular inflammation form of "Uveitis posterior".
  Other Names: Dexamethasone-implant

SUMMARY:
To analyze macula edema formation after cataract surgery called Irvine-Gass-Syndrome.

DETAILED DESCRIPTION:
20 to 25 patients suffering from Irvine Gass Syndrom should be monitored for at least six months, controlled monthly. In all cases best corrected visual acuity, Spectralis-OCT (volume thickness scan), fundus photography (Optomap), intraocular pressure, slitlamp assessment and indirect ophthalmoscopy should be performed on every visit. Fluorescein angiography should be performed at baseline and after 3 and 6 months.

Inclusion criteria:

Patients older than 18 years who develop macula edema secondary to cataract surgery.

- Consent agreement - Patients should be informed that it is possible to get an active medication (Ozurdex implant) as an "on label" indication from the health insurance company if the diagnosis is accepted as an intraocular inflammation form of "Uveitis posterior".

Exclusion criteria:

Visual acuity worse than 20/400, known history of glaucoma and steroid response, any macular disease interfering with visual acuity (DME, AMD, etc.), history of vitrectomy, use of systemic, periocular, or intraocular corticosteroids within 30 days.

Outcome:

* BCVA
* Patients suffering from diabetes mellitus should be evaluated also separately.
* Change in central retinal thickness using optical coherence tomography (OCT)
* Secondary parameters (elevated IOP, retinal detachments, vitreous hemorrhage, endophthalmitis rates)

ELIGIBILITY:
Inclusion Criteria:

Patients older than 18 years who develop macula edema secondary to cataract surgery

Exclusion Criteria:

Visual acuity worse than 20/400, known history of glaucoma and steroid response, any macular disease interfering with visual acuity (DME, AMD, etc.), history of vitrectomy, use of systemic, periocular, or intraocular corticosteroids within 30 days.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 months
  Best corrected visual acuity and visual acuity gain after 6 and 12 months.

SECONDARY OUTCOMES:
Retinal Thickness | 12 months
  Retinal thickness measured by OCT.
Intraocular pressure | 12 months
  Intraocular pressure using Goldmann applanation tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang J Mayer, MD, Principal Investigator — LMU Munich; Christos Haritoglou, MD, PhD, Principal Investigator — LMU Munich
Locations (1):
- Dept. of Ophthalmology, LMU Munich, Munich, Germany